CLINICAL TRIAL: NCT06760507
Title: Evaluating an Evidence-Based Family History Screening Program Adapted to Increase Reach and Uptake of Screening for BRCA-Associated Cancers in Rural Public Health Clinics
Acronym: RSPH5973-23
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Yue Guan, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: STUDY00006068; P30CA138292 (NIH); R37CA276317 (NIH); NCI-2023-05724 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RSPH5973-23 (Other: Emory University)
Record Dates: First submitted 2024-12-18; First posted 2025-01-07 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Ovarian Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aim 2, Arm 1 (Standard Care) (No Intervention): Clinics in the standard care arm follow the existing GA CORE process. Women visiting or calling the clinic are offered FH screening, with public health nurses assisting eligible participants through the GA CORE website. Nurses manually complete data entry using patient identifiers and clinic codes. All referrals are handled manually, and there are no follow-ups for screening-negative results.
- Aim 2, Arm 2 (Adapted Family History Screening Program) (Experimental): The intervention arm includes four key steps designed to enhance the family health screening process. Before the visit, clinics will engage in community outreach using tools such as social media, events, and promotional materials to raise awareness and drive appointment scheduling through the updated GA CORE website 2.0. During the visit, the intervention streamlines the screening process by embedding reminders into workflows and simplifying results communication and documentation. Patients receive theory-based communication materials about their results. After the visit, follow-ups are automated using the updated website 2.0, consolidating data tracking and incorporating risk-stratified communication strategies to encourage appropriate cancer screening behaviors.
  Interventions: Other: Adapted Family History Screening Program

INTERVENTIONS:
Other: Adapted Family History Screening Program — The intervention includes four key steps designed to enhance the family health screening process. Before the visit, clinics will engage in community outreach using tools such as social media, events, and promotional materials to raise awareness and drive appointment scheduling through the updated GA CORE website 2.0. During the visit, the intervention streamlines the screening process by embedding reminders into workflows and simplifying results communication and documentation. Patients receive theory-based communication materials about their results. After the visit, follow-ups are automated using the updated website 2.0, consolidating data tracking and incorporating risk-stratified communication strategies to encourage appropriate cancer screening behaviors.
  Arms: Aim 2, Arm 2 (Adapted Family History Screening Program)

SUMMARY:
This clinical trial adapts and evaluates the effectiveness of a family history screening program (GA CORE) for increasing uptake of genetic screening for BRCA-associated cancers in women who have received care in rural public health clinics in Southwest Georgia. Brief and low-cost family history-based screening assessments to identify families at high risk for BRCA-associated cancers have been endorsed by national guidelines and public health organizations. Georgia is among the few states to have implemented statewide family history screening for BRCA-associated cancers. Despite its potential, current clinic-based approaches that identify at-risk women are not sustainable and show limited reach. Additionally, uptake of follow-up cancer screening is sub-optimal and solely focuses on women screened as high genetic risk. This trial will adapt the existing family history screening program and then evaluate it's effectiveness for increasing the number and diversity of women who receive a history assessment and subsequent access to risk-based services such as genetic counseling and testing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Conduct a multilevel adaptation of GA CORE's existing statewide family history screening program for BRCA-associated cancers to maximize sustainable program reach and improve communication suitability and effectiveness. (Phase I [Exploration & Preparation stages]) II. Use a multi-site, parallel group, cluster randomized controlled trial to evaluate effectiveness of the adapted program relative to the current screening program in promoting uptake of family history screening and correct screening result interpretation among women ages 25 and older who are receiving care in up to 6 of 14 public health clinics in Southwest Georgia. (Phase II [Implementation stage]) III. Use the RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) framework to conduct an implementation research evaluation to measure program process indicators (e.g., reach, fidelity, barriers/facilitators) that may influence program implementation and sustainability. (Phase II [Implementation stage])

OUTLINE:

AIM 1: Participants attend stakeholder advisory committee meetings over 2 hours monthly for 14 months, may attend interviews and/or complete surveys, and attend discussion forums in support of the adaptation of the existing GA CORE screening program on study.

AIM 2: Participating clinics are cluster randomized to 1 of 2 arms.

Standard Care Arm:

Clinics in the standard care arm follow the existing GA CORE process. Women visiting or calling the clinic are offered FH screening, with public health nurses assisting eligible participants through the GA CORE website. Nurses complete data entry manually using patient identifiers and clinic codes. All referrals are done manually, and there are no follow-ups for screening-negative results.

Adapted Intervention Arm:

The intervention arm includes four key steps designed to enhance the family health screening process. Before the visit, clinics will engage in community outreach using tools such as social media, events, and promotional materials to raise awareness and drive appointment scheduling through the updated GA CORE website 2.0. During the visit, the intervention streamlines the screening process by embedding reminders into workflows and simplifying results communication and documentation. Patients receive theory-based communication materials about their results. After the visit, follow-ups are automated using the updated website 2.0, consolidating data tracking and incorporating risk-stratified communication strategies to encourage appropriate cancer screening behaviors.

Positive family history screening results in both arms lead to standard follow-up genetic consultation and testing services.

AIM 3: Participants attend interviews or workshop discussions on study.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1 STAKEHOLDER ADVISORY COMMITTEE: 10 stakeholders representing three constituencies: state cancer control leaders (n=2), participating public health district champions (n=4) (i.e., administrative directors, nurses, clinic staff) and patients (n=4) (i.e., women, age 25 and older who receive their care in the Southwest district)
* AIM 1 DISCUSSION FORUM: 25 years or older
* AIM 1 DISCUSSION FORUM: Women
* AIM 1 DISCUSSION FORUM: English-speaker
* AIM 1 DISCUSSION FORUM: Have completed family history screening during the first 3 months of the project at one of 14 public health clinics in Southwest district
* AIM 1 ORGANIZATIONAL STAKEHOLDER INTERVIEW: Organizational stakeholders (i.e., medical directors, nurses, and clinic staff) at the 14 clinic sites in Southwest district
* AIM 2: Women
* AIM 2: Ages 25 and older
* AIM 2: Who can read English
* AIM 2: Have ever been seen in Women's Health Section through one of participating public health clinics in Southwest district
* AIM 3 POST-INTERVENTION INTERVIEW: Participants from aim 2, regardless of whether they completed the recommended genetic services or not (e.g. complete telegenetic session or genetic testing)
* AIM 3 WORKSHOP DISCUSSION: Medical and administrative directors, nurses, and clinic staff from the six participating clinic sites

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 3209 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Uptake of family history screening | Up to 6 years
  Defined as the number and proportion of the women older than 25 years served by the clinics who complete screening tool. Screening uptake rate at each site will be calculated with a 95% confidence interval. Comparison between arms will be carried out using a mixed-effects logistic regression model.
Screen result interpretation | Up to 6 years
  Will be evaluated by recall of screen result calculated as the concordance of participants' self-reported screen result and their actual result (correct/incorrect) and understanding of the likelihood of carrying a BRCA1/2 mutation (correct/incorrect).

SECONDARY OUTCOMES:
Uptake of genetic consultation and testing | Up to 6 years
  Evaluated as the number and proportion of the women screened as high genetic risk who complete pre-test genetic consultation and testing.
Mammogram screening behaviors | Up to 6 years
  Whether eligible patients underwent mammogram screening (Yes/No).
Acceptance of result validity | Up to 6 years
  Will assess with a scale in which women respond to statements such as, "The information I received about my risk for hereditary breast and ovarian cancer seems accurate"
Emotional processing | Up to 6 years
  Will evaluate cancer fear based utilizing the FHAT questionnaire, a 10-point Likert scale.
Reach | Up to 6 years
  Measured as the number and percentage of eligible women identified based on clinic site records.
Adoption | Up to 6 years
  Measured as the number and percentage of clinic staff who participate in the research project.
Implementation process | Up to 6 years
  The implementation process will be qualitatively assessed to evaluate the perceived acceptability and satisfaction of the adapted program, as well as to identify barriers and facilitators to its delivery and service receipt. At the patient level, we will conduct post-intervention interviews with selected women in the adapted intervention arm. At the organization and provider levels, we will host workshop discussions with organizational implementers of the adapted intervention in late Year 5. During these workshops, we will present the findings of the intervention and gather additional feedback on the program implementation process.
Program sustainability | Up to 6 years
  Evaluated as program potential for sustainability using the Clinical Sustainability Assessment Tool (CSAT) survey.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Guan, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided